CLINICAL TRIAL: NCT03949920
Title: A Prospective Observational Study Investigating the Impact of Migalastat on Cardiovascular Structure and Function in Fabry Disease
Brief Title: A Study of Migalastat in Fabry Disease
Acronym: GALAFAB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B00544; 19/NW/0099 (Other: REC)
Record Dates: First submitted 2019-04-18; First posted 2019-05-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Fabry Disease
Keywords: Fabry; Anderson-Fabry; Migalastat
MeSH Terms: conditions — Fabry Disease | interventions — migalastat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants may agree to donating a blood sample that will be stored in a biorepository for use in future ethically approved research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Migalastat — Participants will be starting Migalastat as part of clinical care. Their initiation onto Migalastat is not determined by this study or it's protocol. Interventions as part of the study will be limited to the study investigations.

SUMMARY:
Fabry disease is a rare metabolic condition characterised by the widespread deposition of sphingolipids in multiple organ systems. Cardiac involvement is common, it occurs in fifty percent of patients and it is the leading cause of death. Despite this, heart and blood vessel (cardiovascular system) manifestations of Fabry disease remain poorly characterised, and it remains unclear which patients benefit from therapy, or when therapy should be initiated. Migalastat is increasingly used to treat fabry disease however the impact of Migalastat on the cardiovascular system is poorly understood. Detailed assessment of the impact of Migalastat on heart and blood vessel structure and function is urgently needed. This observational study will use state of the art, non-invasive investigations to provide greater understanding of the cardiovascular manifestations of Fabry disease and the effects of Migalastat. It will provide insight into which patients respond more effectively to Migalastat, which in turn will facilitate personalisation of therapy, optimisation of the timing of therapy initiation and more cost-effective care.

DETAILED DESCRIPTION:
This is a prospective longitudinal observational study of patients starting Migalastat as part of routine care. Participants will be recruited from outpatient clinics and have a number of investigations before starting therapy and after twelve months of therapy.

Investigations will include a detailed assessment of symptoms and clinical features, blood tests, echocardiography, detailed cardiac MRI scans, heart rhythm monitoring and exercise capacity assessment.

Parameters will be assessed at baseline and at twelve months.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Fabry disease Aged 16 or over Beginning clinical treatment with Migalastat

Exclusion Criteria:

Contraindication to cardiac MRI

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fabry disease commencing Migalastat as part of routine care.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Indexed Left Ventricular Mass (grams/m2) | 12 months
  LV mass, indexed to body surface area, assessed using cardiac MRI.

SECONDARY OUTCOMES:
Change in BSA-indexed LV volumes measured using cardiac MRI, from baseline to 12 months (mls/m2) | 12 months
Change LV ejection fraction, measured using cardiac MRI (%) | 12 months
Change in myocardial extracellular volume, measured using cardiac MRI (%) | 12 months
Change in myocardial tissue T1 and T2 times measured using cardiac MRI (ms) | 12 months
Change in pulmonary artery systolic pressure, measured using echocardiography (mmHg) | 12 months
Change in myocardial PCr/ATP ratio, measured using cardiac MRI spectroscopy (ratio) | 12 months
Change in the number of extra heart beats in a 24 hour period, measured using ambulatory heart monitoring. (number) | 12 months
Change in exercise capacity - Six minute walk test (meters) | 12 months
20. Change in health status (quality of life), measured using change in SF-36 score. (score) | 12 months
Change in Lyso-GB3 blood test levels (nmol/L) | 12 months
Change in Troponin blood test levels (ng/L) | 12 months
Change in NT pro BNP blood test levels (pg/L) | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Manchester University Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.